CLINICAL TRIAL: NCT05696067
Title: Randomized, Double-blind, Placebo-controlled Phase 1/2 Trial of Corfluvec Intranasal Vector Vaccine for the Prevention of COVID-19 in Healthy Volunteers Aged 18 to 60 Years
Brief Title: Evaluation of Corfluvec Vaccine for the Prevention of COVID-19 in Healthy Volunteers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tatyana Zubkova (Other)
Collaborators: MDP-CRO, LLC (Unknown); St. Petersburg State Pavlov Medical University (Other)
Responsible Party: Sponsor-Investigator, Tatyana Zubkova, Head of clinical department, Research Institute of Influenza, Russia
Organization: Research Institute of Influenza, Russia (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KFV-I/II-01/2022
Record Dates: First submitted 2023-01-17; First posted 2023-01-25 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: COVID-19
Keywords: COVID-19; vaccine; influenza vector
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Group 0a (Experimental): Single dose of 7.2 lg EID50 of H3N2 vaccine component
  Interventions: Biological: Corfluvec component 1 low dose
- Group 0b (Experimental): Single dose of 7.5 lg EID50 of H1N1pdm09 vaccine component
  Interventions: Biological: Corfluvec component 2 low dose
- Group 0c (Experimental): Single dose of 8.0 lg EID50 of H3N2 vaccine component
  Interventions: Biological: Corfluvec component 1 high dose
- Group 0d (Experimental): Single dose of 8.3 lg EID50 of H1N1pdm09 vaccine component
  Interventions: Biological: Corfluvec component 2 high dose
- Group 1a (Experimental): Low dose vaccine, two components received three weeks apart
  Interventions: Biological: Corfluvec low dose
- Group 1b (Experimental): High dose vaccine, two components received three weeks apart
  Interventions: Biological: Corfluvec high dose
- Group 1c (Placebo Comparator): Placebo, two doses received three weeks apart
  Interventions: Biological: Placebo
- Group 2a (Experimental): High dose vaccine, two components received three weeks apart
  Interventions: Biological: Corfluvec high dose
- Group 2b (Placebo Comparator): Placebo, two doses received three weeks apart
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Corfluvec component 1 low dose — Participants will receive single intranasal injection of H3N2 recombinant attenuated influenza vector with modified NS gene coding for the N protein fragment of SARS-CoV-2
  Arms: Group 0a
Biological: Corfluvec component 2 low dose — Participants will receive single intranasal injection of H1N1pdm09 recombinant attenuated influenza vector with modified NS gene coding for the N protein fragment of SARS-CoV-2
  Arms: Group 0b
Biological: Corfluvec component 1 high dose — Participants will receive single intranasal injection of H3N2 recombinant attenuated influenza vector with modified NS gene coding for the N protein fragment of SARS-CoV-2
  Arms: Group 0c
Biological: Corfluvec component 2 high dose — Participants will receive single intranasal injection of H1N1pdm09 recombinant attenuated influenza vector with modified NS gene coding for the N protein fragment of SARS-CoV-2
  Arms: Group 0d
Biological: Corfluvec low dose — Participants will receive two intranasal injections of recombinant attenuated influenza vector with modified NS gene coding for the N protein fragment of SARS-CoV-2 tree weeks apart (H3N2 →H1N1pdm09)
  Arms: Group 1a
Biological: Corfluvec high dose — Participants will receive two intranasal injections of recombinant attenuated influenza vector with modified NS gene coding for the N protein fragment of SARS-CoV-2 tree weeks apart (H3N2 →H1N1pdm09)
  Arms: Group 1b; Group 2a
Biological: Placebo — Participants will receive two intranasal injections of placebo three weeks apart
  Arms: Group 1c; Group 2b

SUMMARY:
The aim of the study is to investigate the safety and immunogenicity of a two-component intranasal vaccine for the prevention of COVID-19 in healthy volunteers 18-60 years old

DETAILED DESCRIPTION:
Study include three parts. During the first part the two vaccine components will be administered separately to a small number of seronegative participants in low dose and then high dose to evaluate each component's safety. During the second part vaccine components would be administered one after another with 21 days interval to evaluate safety of the complete vaccine regimen (low dose and high dose). During the third part of the study the high dose vaccine will be administered to participants to evaluate vaccine immunogenicity. The whole study will include 200 participants. Duration of the study for each participant is about 6.5 months (no more than 194 days).

ELIGIBILITY:
Inclusion Criteria:

1. Availability of signed informed consent
2. Adult men and women aged 18-60
3. Diagnosed "healthy" according to the data of standard clinical, laboratory and instrumental examination methods, with the absence of clinically significant changes
4. Body Mass Index (BMI): 18.5≤ BMI ≤30 kg/m2
5. HI antibody titers ≤1:20 to influenza A/H1N1pdm09 and A/H3N2 (only for phase 1)
6. Serum antibodies to the SARS-CoV-2 N-protein not higher than 100 BAU/ml
7. The ability and willingness to make entries in the diary of self-observation, as well as to carry out all the visits foreseen in the study for control medical observation
8. Negative test for alcohol in exhaled air
9. Consent to use effective contraceptive methods throughout their participation in the study
10. Values of the complete blood count and biochemical blood analysis (during the screening) within 0.9*reference range lower limit and 1,1 * reference range upper limit
11. Negative tests for HIV, hepatitis B, hepatitis C, and syphilis

Exclusion Criteria:

1. Contact with COVID-19 patients within 14 days prior to the start of the clinical study
2. Positive rapid test result for SARS-CoV-2 antigen
3. Participation in another clinical study within three months prior to the start of the current study; planning to participate in another study during the current study period.
4. Immunization with any other non-study vaccine product, including COVID-19 vaccination within four weeks prior to enrollment in the current study, or refusal to postpone such until the end of the four-week period after completion of the current study
5. Regular use of nasal irrigation therapy during the last six months prior to enrollment in the current study or episodic use of the above method of treatment in the two weeks prior to the screening
6. History of frequent nosebleeds (>5) during the year prior to the current study
7. Clinically significant anatomic pathology or the presence of surgical intervention in the sinus area, paranasal sinuses, or traumatic injuries of the nose within a month before screening
8. Symptoms of acute respiratory disease, including fever, or other acute illness at the time of screening or within two weeks prior to screening
9. Treatment with immunoglobulins or other blood derived medications in the three months prior to screening or planning such treatment during the period of participation in the current study; donation of blood/plasma (450 ml or more) less than 2 months prior to screening
10. The presence or suspicion of the presence of various immunosuppressive or immunodeficiency conditions or continuous use (the drug was prescribed for more than 14 days without a break) of immunosuppressive drugs, immunomodulators for 6 months before the screening
11. History of bronchial asthma
12. Hypersensitivity and the presence of severe allergic reactions, including Quincke's edema, anaphylactic shock after the previous administration of any vaccine
13. History of wheezing after previous immunization with live influenza vaccine
14. Other adverse events after immunization (fever above 40°C, syncope, non-febrile convulsions, anaphylaxis) when there is a minimal likelihood that they are associated with a previous administration of any vaccine
15. Suspicion of hypersensitivity to any component of the study vaccine, including egg protein
16. Seasonal (in spring or autumn) increased sensitivity to the effects of natural factors
17. Acute or chronic clinically significant lung, cardiovascular, hepatic, endocrine, neurological, or psychiatric disorders, or impaired renal function identified by history, physical examination, or clinical laboratory findings that, in the opinion of the investigator, may influence the outcome of the study
18. History of leukemia or any other malignant diseases of the blood or solid malignant neoplasms of other organs
19. History of thrombocytopenic purpura or bleeding disorders
20. History of convulsions
21. The presence or suspicion of the presence of various immunosuppressive or immunodeficiency conditions, including HIV infection
22. Tuberculosis or residual changes after tuberculosis according to the anamnesis and / or available medical documentation
23. Chronic alcohol dependence or chronic use of illicit drugs, drug abuse
24. Claustrophobia and social phobia according to history and / or available medical records
25. For women of reproductive age - lactation, pregnancy or suspected pregnancy, early postpartum period
26. Premenopausal women (last menstrual period <1 year prior to signing informed consent) who are not surgically sterile and women who are of reproductive potential but do not use or plan to use valid birth control throughout the study and do not agree to perform a urine pregnancy test while participating in the study
27. Military personnel undergoing military service on conscription
28. Persons in custody in pre-trial detention centers and serving sentences in places of deprivation of liberty
29. Special diet (eg, vegetarian, vegan, salt-restricted) or lifestyle (night work, extreme physical activity)
30. Any condition that, in the opinion of the investigator, may increase the risk to the health of a volunteer participating in the study or affect the results of the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with local and systemic adverse events (AEs) and serious adverse events (SAEs) | Throughout the study, average of 6.5 months
  Number of participants with AEs and SAEs including those of particular interest:
  * immediate AEs (allergic reactions) occurring within 2 h after vaccination;
  * post-vaccination reactions between 2 h and a subsequent 7 days;
  * other AEs including unexpected clinical manifestations of a local and systemic nature occurring on the day of vaccination and the following 7 days;
  * deviations of laboratory parameters of analyzes of blood and urine samples and data from instrumental studies (ECG) obtained on Days 3, 7, 23 and 27;
  * all SAEs occurring up to 3 weeks after each vaccination; late AEs occurring after study Day 42 through Day 180±5;
  * influenza A virus shedding detected by rapid test in nasal swab samples
Level of SARS-CoV-2 antigen specific cytokine producing T-cells | Throughout the 42±2 study days
  Change from baseline in the level of cytokine producing T-cells upon in vitro stimulation of PBMC with SARS-CoV-2 N protein peptide epitopes measured by ICS/ELISPOT
Level of SARS-CoV-2 antigen specific cytokine release in whole blood assay | Throughout the 42±2 study days
  Change from baseline in the cytokine concentration in whole-blood cytokine release assay upon in vitro stimulation with SARS-CoV-2 N protein peptide epitopes
Level of SARS-CoV-2 antigen specific mucosal and systemic IgA and IgG antibody | Throughout the 42±2 study days
  Change from baseline in the levels of IgA and IgG antibody to SARS-CoV-2 N protein measured in ELISA in saliva/nasal secret and serum

SECONDARY OUTCOMES:
Number of responders to vaccination according to the fold increase in the level of specific T-cell response | Days 7, 21, 27, 42±2
  Proportion of participants exhibiting significant increase in the level of specific T-cell response to SARS-CoV-2 N protein after vaccination in comparison to baseline. The increase in the parameter is considered significant if it exceeds the specified range, which is a 95% CI for mean value of parameter fold change in the Placebo group at assessment day compared to Day 1
Seroconversion rate of SARS-CoV-2 antigen specific antibody | Days 21, 42±2
  Proportion of participants who have at least a 4-fold increase in post-vaccination antibody titers in comparison to baseline

OTHER OUTCOMES:
Concentration of cytokines in nasal secrets after vaccination | Throughout the first 48h of the study
  Change from the baseline in the concentration of cytokines in nasal secrets measured in ELISA/Multiplex system
Influenza specific local and systemic antibody immune response | Throughout the 42±2 study days
  Change from baseline in the uiters of influenza specific antibodies in serum and saliva/nasal secret measured in ELISA, HI, MNA and corresponding seroconversion rates.
SARS-CoV-2 and influenza specific antibody and T-cell immune response (follow-up) | Days 90±3, 180±5
  Specific systemic antibody and T-cell immune response to SARS-CoV-2 N protein and influenza viruses (A/H1N1pdm09, A/H3N2) measured in ELISA, ISC/ELISPOT, whole-blood cytokine release assay.
Efficacy against symptomatic COVID-19 and influenza | Throughout the study, average of 6.5 months
  Number of laboratory-confirmed symptomatic cases of COVID-19 and influenza

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - Pavlov First State Medical University of St. Petersburg, Saint Petersburg
  - Smorodintsev Research Institute of Influenza, Saint Petersburg